CLINICAL TRIAL: NCT04244409
Title: INvestigational Study Into Transplantation of the Uterus
Acronym: INSITU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Womb Transplant UK (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Ben Jones, Principal Investigator, Imperial College Healthcare NHS Trust
Other Study IDs: WombTransplantUK
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Mayer-Rokitansky-Kuster Syndrome; Asherson's Syndrome; Postpartum Hemorrhage; Cervical Cancer
Keywords: Gynaecology; Immunosuppression; In-vitro Fertilisation; Infertility; MRKH; Pregnancy; Transplantation; Uterus
MeSH Terms: conditions — Mullerian aplasia; Postpartum Hemorrhage; Uterine Cervical Neoplasms; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study on cohort of 10 women undergoing uterine transplantation using deceased donors

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age - 24-38 (or 40 if eggs frozen <38)
3. AUFI

   1. Normal length vagina
   2. No renal pathology
4. BMI <30kg/m2
5. ASA grade I
6. Meet psychological criteria
7. Meet HFEA criteria for IVF
8. Eligible for NHS treatment
9. Speak fluent English

Exclusion Criteria:

1. Unsuccessful oocyte retrieval (<10 good quality embryos)
2. Previous multiple/significant surgeries
3. Severe endometriosis
4. Cancer patients <5 years in remission
5. Previous living childbirth, adopted child or child born through surrogacy
6. HIV or Hepatitis B / C positive
7. Skin or intestinal neovagina

Ages: 24 Years to 38 Years | Sex: Female
Age Groups: Adult
Study Population: Women with absolute uterine factor infertility
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-02-18 (Estimated); Study Completion 2024-02-18 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 5 years

SECONDARY OUTCOMES:
Pregnancy rate | 5 years
Transplant success rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Hospital, Imperial College NHS Trust, London, United Kingdom